CLINICAL TRIAL: NCT00930813
Title: A Prospective, Multicenter, Single Blind, Randomized, Controlled Trial Comparing the Lutonix Catheter vs. Standard Balloon Angioplasty for Treatment of Femoropopliteal Arteries With and Without Stenting.
Brief Title: LEVANT I, The Lutonix Paclitaxel-Coated Balloon for the Prevention of Femoropopliteal Restenosis
Acronym: LEVANT I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL0012-01
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Atherosclerosis; Vascular Disease; Arteriosclerosis
Keywords: Drug coated balloon; SFA disease; Femoropopliteal disease; Angioplasty; PAD; Paclitaxel; Tubulin modulators; Antineoplastic Agents; Mitosis Modulators; Balloon angioplasty; Local drug delivery; Restenosis; Drug-coated balloon
MeSH Terms: conditions — Atherosclerosis; Vascular Diseases; Arteriosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lutonix Catheter (Experimental): Paclitaxel coated Balloon Catheter
  Interventions: Device: Lutonix Catheter
- Standard uncoated Balloon Angioplasty Catheter (Active Comparator): uncoated angioplasty balloon
  Interventions: Device: Standard uncoated Balloon Angioplasty Catheter

INTERVENTIONS:
Device: Lutonix Catheter — Paclitaxel Coated Balloon Catheter
  Other Names: DCB; Drug coated balloon
  Arms: Lutonix Catheter
Device: Standard uncoated Balloon Angioplasty Catheter — plain, uncoated angioplasty balloon catheter
  Arms: Standard uncoated Balloon Angioplasty Catheter

SUMMARY:
The purpose of the study is to assess the safety and efficacy of the Lutonix Catheter for treatment of stenosis of the femoropopliteal arteries by direct comparison to standard balloon angioplasty.

DETAILED DESCRIPTION:
The LEVANT I trial will enroll patients presenting with clinical evidence of claudication or critical limb ischemia and an angiographically significant lesion in the femoropopliteal arteries. Patients will be randomized to treatment with either the Lutonix Catheter or standard balloon angioplasty after predilation.

ELIGIBILITY:
Inclusion Criteria:

Clinical Criteria

* Male or non-pregnant female ≥18 years of age.
* Rutherford Clinical Category 2-5
* Patient is willing to provide informed consent and comply with the required follow up visits, testing schedule, and medication regimen Angiographic Criteria
* A single de novo or restenotic atherosclerotic lesion >70% in the SFA or popliteal artery that is ≥4 cm and ≤15 cm in total length.
* Reference vessel diameter ≥4 mm and ≤ 6mm
* Successful wire crossing of lesion
* A patent inflow artery free from significant lesion (>50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of inflow artery lesions)

Exclusion Criteria:

* Pregnant or planning on becoming pregnant in < 2yrs
* Live expectancy of <2 years
* Patient actively participating in another investigational device or drug study
* History of hemorrhagic stroke within 3 months
* Previous or planned surgical or interventional procedure within 30 days of index procedure
* Chronic renal insufficiency with creatinine >2.5 mg/L
* Prior surgery of the target lesion
* Inability to take required study medications
* Anticipated use of IIb/IIIa inhibitor prior to randomization
* Lesion length is <4 cm or >15 cm or there is no normal proximal arterial segment in which duplex ultrasound velocity ratios can be measured
* Known inadequate distal outflow
* Significant inflow disease
* Acute or sub-acute thrombus in target vessel
* Severe lesion calcification
* Acute vessel occlusion or sudden symptom onset
* Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, etc.)
* Prior participation in the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Sint Blasius, Dendermonde, Belgium
- Germany (9):
  - Herz Zentrum, Bad Krozingen
  - Jewish Hospital, Berlin
  - St Katharenen Cardiovascular Center, Frankfurt
  - Hamburg Unversity Cardiovascular Center, Hamburg
  - Park Krankenhaus - University of Leipzig, Leipzig
  - Universitätsklinikum, Magdeburg
  - St. Franziskus, Münster
  - Klinikum Rosenheim, Rosenheim
  - Katharinenhospital, Stuttgart

REFERENCES:
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Derived] Ouriel K, Adelman MA, Rosenfield K, Scheinert D, Brodmann M, Pena C, Geraghty P, Lee A, White R, Clair DG. Safety of Paclitaxel-Coated Balloon Angioplasty for Femoropopliteal Peripheral Artery Disease. JACC Cardiovasc Interv. 2019 Dec 23;12(24):2515-2524. doi: 10.1016/j.jcin.2019.08.025. Epub 2019 Sep 28. PMID 31575518
- [Derived] Scheinert D, Duda S, Zeller T, Krankenberg H, Ricke J, Bosiers M, Tepe G, Naisbitt S, Rosenfield K. The LEVANT I (Lutonix paclitaxel-coated balloon for the prevention of femoropopliteal restenosis) trial for femoropopliteal revascularization: first-in-human randomized trial of low-dose drug-coated balloon versus uncoated balloon angioplasty. JACC Cardiovasc Interv. 2014 Jan;7(1):10-9. doi: 10.1016/j.jcin.2013.05.022. PMID 24456716

RESULTS

PARTICIPANT FLOW:
Groups:
- Lutonix DCB Catheter: Lutonix DCB: Paclitaxel Coated Balloon Catheter
- Uncoated PTA Balloon Catheter: Standard, uncoated, off-the-shelf PTA Balloon Angioplasty Catheter
Period: Overall Study
Arm/Group | Lutonix DCB Catheter | Uncoated PTA Balloon Catheter
Started | 49 | 52
Completed | 41 | 38
Not Completed | 8 | 14
Not completed — Death | 4 | 5
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix Catheter | Standard Uncoated Balloon Angioplasty Catheter | Total
Number analyzed (Participants) | 49 | 52 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 70 (10) | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 34 | 30 | 64
Lesion location [Number; unit: participants]
  SFA | 45 | 49 | 94
  Popliteal | 4 | 3 | 7
Lesion Length [Mean (Standard Deviation); unit: mm] | 81 (37) | 80 (38) | 81 (38)
Lesion totally occluded [Number; unit: participants]
  Yes | 20 | 22 | 42
  No | 29 | 30 | 59
Rutherford Class [Number; unit: participants]
  2 (Moderate claudication) | 11 | 11 | 22
  3 (Severe claudication) | 35 | 37 | 72
  4 (Ischemia rest pain) | 1 | 2 | 3
  5 (Minor tissue loss) | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Angiographic Late Lumen Loss
Description: Loss in analysis segment (the treated segment including 10mm distal and proximal) minimal lumen diameter from post-procedure through follow-up angiography at 6 months.
Time Frame: 6 months
Population: Intent-to-treat among completers, including all patients with valid angiographic imaging analyzable by the core lab.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Lutonix DCB Catheter: Lutonix Paclitaxel Coated Balloon Catheter
- Standard Uncoated PTA Catheter: Standard off-the-shelf uncoated PTA Catheter
Arm/Group | Lutonix DCB Catheter | Standard Uncoated PTA Catheter
Number analyzed (Participants) | 39 | 35
mm | 0.46 (1.13) | 1.09 (1.07)
Statistical Analysis 1: Comparison: Lutonix DCB Catheter vs Standard Uncoated PTA Catheter; The study required 100 subjects to provide 80% power to detect a clinically meaningful difference in late lumen loss of 15% of reference vessel diameter between treatment groups on the basis of a 2-sample Student t test with 2-sided alpha 0.05; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

2. Secondary Outcome: Safety - Device Related Adverse Events
Time Frame: 30 days
Population: ITT
Measure: Number; unit: participants
Arm/Group | Lutonix DCB Catheter | Uncoated PTA Balloon Catheter
Number analyzed (Participants) | 49 | 52
participants | 0 | 4

3. Secondary Outcome: Primary Patency of Treated Segment
Time Frame: 6, 12, 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Target Lesion Revascularization
Time Frame: 6, 12, 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Target Vessel Revascularization
Time Frame: 6, 12, 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Device Success
Description: Successful delivery and deployment of the first inserted study device (in overlapping setting a successful delivery and deployment of the first and second study device) at the intended target lesion and successful withdrawal of the study device with attainment of final residual stenosis of less than 30% of the target lesion by quantitative vessel angiography (QVA).
Time Frame: at procedure
Reporting Status: Not Posted

7. Secondary Outcome: Procedural Success
Description: Completion of the procedure with less than 30% residual stenosis by QVA of the target lesion (after prolonged dilation and stenting, if necessary)
Time Frame: at procedure
Reporting Status: Not Posted

8. Secondary Outcome: Change in Ankle-brachial Index
Time Frame: pre-procedure, 6, 12 and 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ)
Time Frame: pre-procedure, 6, 12 and 24 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in Rutherford Grade
Time Frame: pre-procedure,6, 12 and 24 months
Reporting Status: Not Posted

11. Secondary Outcome: Serum Paclitaxel Levels - in Subsets of Patients
Time Frame: 0, 1, 3 hours and pre-discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Lutonix Catheter | Standard Uncoated Balloon Angioplasty Catheter
Serious Adverse Events (participants affected / at risk) | 39/49 | 39/52
Other Adverse Events (participants affected / at risk) | 17/49 | 28/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Catheter (N=49) | Standard Uncoated Balloon Angioplasty Catheter (N=52)
Target lesion - Restinosis (Vascular disorders) | 13 (20) | 17 (22)
Abscess (General disorders) | 1 (1) | 0 (0)
Access site complication: pseudo aneurysm (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Amputation (Surgical and medical procedures) | 1 (6) | 1 (1)
Angina, stable (Cardiac disorders) | 3 (3) | 2 (3)
Arrhythmia - Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - Other (Cardiac disorders) | 1 (1) | 2 (2)
Arrhytmia - Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Battery depletion of pacemaker (General disorders) | 1 (1) | 0 (0)
Bleeding out of mouth and nose (General disorders) | 1 (1) | 0 (0)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Death (Cardiovascular) (Vascular disorders) | 1 (1) | 1 (1)
Death (non-cardiac or neurological) (General disorders) | 1 (1) | 1 (1)
Diffuse bleeding on metatarsus (General disorders) | 1 (1) | 0 (0)
Fracture (bone) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal: other infectious / inflammatory (Gastrointestinal disorders) | 1 (1) | 0 (0)
Groin hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Renal and urinary disorders) | 1 (1) | 1 (1)
Malfunction of the defibrillator (General disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Not any healing of ulceration on right foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Patient fell down, pain in the back (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patient was injured during fall : bruise left hip (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Persistent wound healing disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Stroke - ischemic (Cardiac disorders) | 2 (2) | 0 (0)
Target vessel - Restenosis (Vascular disorders) | 2 (2) | 2 (3)
TIA (Cardiac disorders) | 1 (1) | 0 (0)
Vessel specific complication (not puncture site or target vessel): Arterial occlusion (Vascular disorders) | 4 (4) | 6 (7)
Vessel specific complication (not puncture site or target vessel): Arterial thrombosis (Vascular disorders) | 1 (1) | 2 (3)
Vessel specific complication (not puncture site or target vessel): Atherosclerosis (Vascular disorders) | 5 (6) | 14 (18)
Vessel specific complication (not puncture site or target vessel): Embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vessel specific complication (not puncture site or target vessel): Restenosis (Vascular disorders) | 9 (10) | 7 (9)
Worseness of ulceration on amputation wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence after CABG (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound infection after amputation of second toe (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Access site complication: Arterial occlusion puncture site (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Aggregate change of pacemaker (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arthralgia (Infections and infestations) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Claudication (Vascular disorders) | 0 (0) | 2 (2)
Colon carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Control coronary angiography (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Defibrillator control (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dementia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness / vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fall from bed - urinary bladder infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Local infection (Infections and infestations) | 0 (0) | 2 (3)
Target lesion - Occlusion / closure (Vascular disorders) | 0 (0) | 3 (4)
Vessel specific complication (not puncture site or target vessel): Hematoma / bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound lower leg with infection (MRSA) and maggots (Infections and infestations) | 0 (0) | 1 (1)
Target lesion - Thrombus - in-lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Catheter (N=49) | Standard Uncoated Balloon Angioplasty Catheter (N=52)
Access site complication: pseudo aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Access site complication: Hematoma/bleeding puncture site (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Claudication (Vascular disorders) | 4 (4) | 4 (4)
Hypertension (Renal and urinary disorders) | 0 (0) | 3 (3)
Target lesion - Dissection (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Target lesion - Restenosis (Vascular disorders) | 7 (11) | 4 (4)
Vessel specific complication (not puncture site or target vessel): Atherosclerosis (Vascular disorders) | 1 (1) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days